CLINICAL TRIAL: NCT01996592
Title: Novel Approach Using Pre-surgery Psychosocial State and Pain Trajectory Methods to Identify Patient Characteristics and Predict Patients at Risk for Persistent Pain After Cesarean Delivery
Brief Title: Persistent Pain After CS Delivery
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00022468
Record Dates: First submitted 2013-11-21; First posted 2013-11-27 (Estimated); Results first posted 2018-08-13 (Actual); Last update posted 2018-08-13 (Actual); Status verified 2018-08

CONDITIONS: Persistent Pain After Delivery
Keywords: chronic pain; cesarean section pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- cesarean section deliveries: those subjects having an elective cesarean section will complete an informed consent form, complete the preoperative questionnaire, and then be contacted for 60 days postoperatively

SUMMARY:
Many factors influence the development of persistent pain after CS (chronic pain) as well as post-partum depression. We are attempting to use trajectory pain methods in an attempt to identify those at risk for the development of persistent pain post delivery using a daily method of contact for the determination of pain scores. Assessments are also done evaluating satisfaction of pain management and maternal/infant bonding opportunities. Physical activity is monitored by subject's wearing a Fitbit with correlation being done with pain scores obtained over 60 days postop with eligible subjects..

DETAILED DESCRIPTION:
Subjects are contacted on a daily basis after having a cesarean delivery to determine current pain, current pain unpleasantness, worst pain, worst pain unpleasantness, average pain, and average pain unpleaseantness. Preoperatively subjects complete a psycho-social/depressive screening questionnaire. Pain treatments/satisfaction assessments are captured for the first 24 hours. Mother/baby outcomes are also captured. Physical activity and pain scores are also correlated with the subject's wearing of a Fitbit physical activity bracelet with eligible subjects for 60 days post-delivery.

ELIGIBILITY:
Inclusion Criteria:

* >/= 18 years of age English speaking

Exclusion Criteria:

non-English speaking

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: those subjects who are scheduled to have an elective cesarean section (CS) and able to complete a preoperative psychosocial/depressive questionnaire and who agree to be contacted on a daily basis for 60 days postoperatively
Sampling Method: Probability Sample
Enrollment: 575 (Actual)
Dates: Start 2013-05; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Booth, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Forsyth Medical Center, Winston-Salem, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Elective cesarean section patients >/= 18 years of age who agree to be contacted for 8 weeks after delivery to obtain pain scores
Period: Overall Study
Arm/Group | Cesarean Section Deliveries
Started | 575
Completed | 530
Not Completed | 45
Not completed — no response to text/no diary entry | 32
Not completed — change in surgical date | 4
Not completed — Withdrawal by Subject | 5
Not completed — change in mode of delivery | 4

BASELINE CHARACTERISTICS:
Arm/Group | Cesarean Section Deliveries
Number analyzed (Participants) | 530
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 530
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 575 enrolled; 530 analyzed. 45 subjects were excluded for the following reasons: no response to text/no diary entry: 32 change in surgical date: 4 withdrew consent prior to study initiation: 5 change in mode of delivery: 4
  Participants
    Female | 530
    Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: 575 enrolled; 530 analyzed. 45 subjects were excluded for the following reasons: no response to text/no diary entry: 32 change in surgical date: 4 withdrew consent prior to study initiation: 5 change in mode of delivery: 4
  Participants
    American Indian or Alaska Native | 0
    Asian | 3
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 138
    White | 384
    More than one race | 0
    Unknown or Not Reported | 5

OUTCOME MEASURES:

1. Primary Outcome: Persistent Pain-PERCEIVED STRESS Scores Stratified by the Rate of Recovery
Description: By identifying preoperative risk factors for chronic pain and mapping out the trajectory of pain after cesarean delivery, we may be able to use novel pharmacologic or psychological interventions to alter postoperative pain trajectories. Two predominant risk factors have been determined thus far to put those at risk. They are emotional distress/depression and perceived stress. The 530 participants recovery pain scores were broken down into 3 subgroups--group 1 is those who had the fastest recovery, group 2 which is the "average" recovery, and group 3 which is the group with the slowest recovery.
Time Frame: 60 days
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Group 1-perceived Stress Scores: Subjects who had the fastest recovery
- Group 2 Perceived Stress Scale: Subjects who experienced average recovery
- Group 3 Perceived Stress Scale: Subjects who experienced the slowest recovery from surgery
Arm/Group | Group 1-perceived Stress Scores | Group 2 Perceived Stress Scale | Group 3 Perceived Stress Scale
Number analyzed (Participants) | 307 | 170 | 53
units on a scale | 11.4 (5.8) | 12.9 (5.8) | 15.4 (5.4)
Statistical Analysis 1: Comparison: Group 1-perceived Stress Scores; PROMIS -perceived stress scale was utilized (a validated test). Scoring ranges from 0-40, with the following ranges indicative of low, moderate, or high perceived stress: 0-13=low stress 14-26=moderate stress 27-40=high perceived stress; Test type: Other; p < 0.01, ANOVA — p-value was calculated

2. Primary Outcome: Persistent Pain-EMOTIONAL DISTRESS
Description: By identifying preoperative risk factors for chronic pain and mapping out the trajectory of pain after cesarean delivery, we may be able to use novel pharmacologic or psychological interventions to alter postoperative pain trajectories. Two predominant risk factors have been determined thus far to put those at risk. They are emotional distress/depression and perceived stress. The 530 participants recovery pain scores were broken down into 3 subgroups--group 1 is those who had the fastest recovery, group 2 which is the "average" recovery, and group 3 which is the group with the slowest recovery.
  PROMIS Emotional Distress-Depression Short form utilized for this outcome. scoring for this ranges from 8-40, with the higher the score the worse the distress
Time Frame: 60 days
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Group 1-emotional Distress Scores: Subjects who had the fastest recovery
- Group 2 Emotional Distress Scale: Subjects who experienced average recovery
- Group 3 Emotional Distress Scale: Subjects who experienced the slowest recovery from surgery
Arm/Group | Group 1-emotional Distress Scores | Group 2 Emotional Distress Scale | Group 3 Emotional Distress Scale
Number analyzed (Participants) | 307 | 170 | 53
units on a scale | 10.7 (3.8) | 11.5 (4.2) | 12.8 (4.5)
Statistical Analysis 1: Comparison: Group 1-emotional Distress Scores vs Group 2 Emotional Distress Scale vs Group 3 Emotional Distress Scale; Test type: Other; p < 0.01, ANOVA — p-value was calculated

ADVERSE EVENTS:
Arm/Group | Cesarean Section Deliveries
All-Cause Mortality (participants affected / at risk) | 0/530
Serious Adverse Events (participants affected / at risk) | 0/530
Other Adverse Events (participants affected / at risk) | 0/530

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes